# A Randomized controlled trial of 2% chlorhexidine gluconate skin preparation cloths for the prevention of post op surgical site infections in spine patients

November 1, 2018

NCT02490631

# **Protocol Title**

A Randomized controlled trial of 2% chlorhexidine gluconate skin preparation cloths for the prevention of post op surgical site infections in spine patients

Elizabeth Card, MSN, APN, FNP-BC, CPAN, CCRP. Research Nurse Practitioner: Anesthesiology



Sub Investigators
Joseph Cheng, MD
Damon Michaels, BS, CCRP
Steve Klintworth, RN
Edward Sherwood, MD, PhD
Gail Mayo, RN, CCRP
Nancy Wells, DNSc, RN

# Confidential

Department of Anesthesiology Vanderbilt University

# **Protocol Title**

A Randomized controlled trial of 2% chlorhexidine gluconate skin preparation cloths for the prevention of post op surgical site infections in spine patients

Elizabeth Card, MSN, APN, FNP-BC, CPAN, CCRP. Research Nurse Practitioner: Anesthesiology



Sub Investigators
Joseph Cheng, MD
Damon Michaels, BS, CCRP
Steve Klintworth, RN
Edward Sherwood, MD, PhD
Gail Mayo, RN, CCRP
Nancy Wells, DNSc, RN

# Confidential

Department of Anesthesiology Vanderbilt University

# Table of Contents:

- 1. Background and Significance
- 2. Hypothesis
- 3. Study Objectives
- 4. Methods
- 5. Patient Population
- 6. Enrollment
- 7. Inclusion/Exclusion Criteria
- 8. Data Collection
- 9. Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others:
- 10. Statistical Plan
- 11. Privacy/Confidentiality Issues
- 12. Follow-up and Record Retention

# 1. Background and Significance:

Surgical site infection (SSI) following spinal surgery is a frequent complication and results in higher morbidity, mortality and healthcare costs. SSI following adult spinal surgery is a frequent complication that has been reported to occur in 0.7–12.0% of patients and result in higher postoperative morbidity, mortality and health care costs. Vanderbilt University Medical Center SSI rate is 7%. Treatment for SSI can be challenging often requiring revision surgery, long-term antibiotics, and prolonged hospitalization. The accurate identification of risk factors is thus important in the development of strategies to prevent these potentially devastating infections.

The New CDC-definitions for surveillance of surgical site infections (1992) take into account 3 classes of surgical site infections (SSI): superficial incisional SSI, deep incisional SSI, and organ/space SSI. The most prevalent host-related risk factors for development of SSI are advanced age, morbid obesity, disease severity, an ASA score > 2, prolonged preoperative hospital stay, and infection at distal sites. Microbial contamination of the surgical site occurs mainly during the surgical intervention.

Although exogenous contamination from the surgical suite may be of concern, especially in clean operations, most surgical site infections are caused by microorganisms of the patient's own skin flora. SSI rates vary according to the type and duration of the surgical procedure. Proper surgical technique is probably the most important factor in the prevention of SSI. Modification of patient risk factors should be attempted whenever possible through use of

Modification of patient risk factors should be attempted whenever possible through use of adequate protocols for antimicrobial prophylaxis with antibiotics should be followed. Routine surveillance of surgical site infections is beneficial for SSI prevention and early detection. Additional prevention aimed at decreasing number of microorganisims on patient's skin preoperatively may decrease rates of SSI. Prior studies have reported daily use of 2% chlorhexidine gluconate (CHG) cloths has decreased rates of nosocomial bloodstream infections in those with central line catheters. Another study reported decreasing SSIs up to 50% when nursing staff instituted utilization of CHG cloths pre-op and daily post-op cleansing in-hospital. However, use of CHG cloths pre-operatively has not been routinely instituted. Many hospitals and service lines do not have a protocol for their use. Therefore study of such a population may prove worthy, as currently VUMC neuro-spine patients do not routinely utilize preoperative skin cleansing with CHG cloths.

This study proposes a randomized, controlled trial of neuro-spine patients of 2% chlorhexidine gluconate skin preparation cloths for the prevention of post op surgical site infections in spine patients.

# 2. Hypothesis:

Use of CHG cloths the night before and morning of surgery (neckline to toes) will affect (decrease rates) of SSI compared to patients who receive routine standard of care (soap and water pre-op, day of surgery and daily post-operative).

# 3. Study Objectives:

- Randomize consented patients pre-operative to either study group (of 2% chlorhexidine gluconate cloths the night before and morning of surgery) or control (standard of care cleansing with soap and water) with follow-up through discharge for evaluation of SSI
- Evaluation for SSI development at 6 week (+/-) 1 week post-op visit.

 Measure change in skin flora by comparing skin swab cultures of those using the cloths and those who do not on day of surgery, post-op day 4 or hospital discharge and postop day 30

#### Methods:

Pre-operatively patients scheduled for neurosurgical spine cases will be evaluated and approached for interest, if consenting process completed, patients will be randomized to one of 2 arms in 1:1 through a block randomization table.

Those enrolled into the study arm will receive the CHG cloths and instructions for use from research personal. Those randomized to the control arm will receive standard of care skin cleansing by nursing staff.

All subjects who have signed consent will have a skin swab culture taken the day of screening and prior to cleansing with Chlorhexidine gluconate wipes close to the intended incision line. We will also obtain skin swab cultures at site of incision preoperatively on the day of surgery, post-op day 4 or time of discharge (which ever comes first) and at the 30 day follow up.

Both groups will be evaluated daily by study personnel for the development of SSI until postop day 4 or hospital discharge whichever one comes first.. Additional evaluations will take place at the 30 day (+/- 7 days) post-op visit. Blinded evaluators utilizing the CDC guideline will grade the incision line for presence of SSI. Measured change in skin flora will be performed by comparing skin swab cultures of intervention group versus standard of care group and individual changes pre and post operatively.

# 5. Patient Population:

Neurosurgical spine patients at Vanderbilt University Medical Center

#### 6. Enrollment:

170 patients will be enrolled.

# 7. Inclusion/Exclusion Criteria:

#### Inclusion Criteria

Patients scheduled for a neuro-spine procedure and have 2 of the following risk factors: Diabetic OR BMI>30 OR ASA>2 OR pre-operatively hospitalized OR >60 years old OR chronic steroids/immunosuppressive medications OR prior history of SSI

#### **Exclusion Criteria**

- 1) Unable to consent
- 2) Non English speaking
- 3) Known allergy to any of the ingredients contained in SAGE chlorhexidine gluconate cloths
- 4) Current infection or history of spine infections.
- 5) Patients with tumors or intradural spinal pathology.

# 8. Data Collection:

Data regarding demographics, health history and status, surgical course and hospitalization will be collected and entered into an electronic database. Patient data will be de-identified once entered into the database. Shared data will always be de-identified and accessed through Redcap, a secure web-based system.

# 9. Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others:

Events determined by the Principal Investigator (PI) to be unanticipated problems involving risks to subjects will be reported by the PI or sub-investigator to the IRB within 10 working days of the Investigator's knowledge of the problem.

#### 10. Statistical Plan:

We are planning a study of independent cases and controls with 1 control(s) per case. Prior data indicate the rate of infection in the control group (those with risk factors, including superficial SSI) is 0.5, then just 150 evaluable subjects are needed to detect a 50% or greater reduction, with 80% power. We can also design a statistical analysis plan that uses the grade of SSI instead of binary yes/no to indicate presence of SSI. This should increase the power as well, for instance, if the SAGE cloths reduce the severity of (but does not completely prevent) infection in some patients.

# 11. Privacy/Confidentiality Issues

All reasonable efforts will be made to keep a patient's protected health information (PHI) private and confidential. There will be limited access to electronic medical records and deidentification of all records. Federal privacy guidelines will be followed when using or sharing any protected health information.

Data will be stored in Redcap, a secure web-based database conforming to the latest Vanderbilt IS security policies. Data from the study will be reported only in the aggregate.

Under the supervision of each site's PI, Vanderbilt research team members will view research records and collect data as identified above. Medical records will be stored separately from the data and remain on-site. All de-identified data-points will be entered directly into Redcap, a secure web-based database. No identified information will leave the site.

All study staff have completed employee education regarding patient confidentiality and have completed Human Subjects protection education (CITI course) as specified by the Vanderbilt IRB.

Through these interventions, we expect risks to privacy to be minimized.

# 12. Follow-up and Record Retention

Research Records will be retained by the Nursing Research Office for a period of six (6) years after the submission of the final report and close-out procedures on the research project for which the Research Records were prepared.

The retention of the original Research Records shall be the responsibilityNursing Research Office .

# Study Schema

| Procedure | screening | Day of surgery | POD 1 | POD 2 | POD 3 | POD4 or<br>discharge | 6 weeks<br>± 1 week<br>follow up<br>visit |
|---|---|---|---|---|---|---|---|
| Written informed consent | X | | | | | | |
| Medical history | Х | | | | | | |
| Urine pregnancy test | | Х | | | | | |
| BMI | Х | | | | | | |
| Vital signs (HR, RR,<br>BP, T) | X | Х | X | X | X | x | Х |
| Randomization | Х | | | | | | |
| SAGE cloths for<br>treatment arm <sup>1</sup> | X | Х | | | | | |
| Standard of care;<br>soap and water for<br>control arm | х | х | х | х | х | X | |
| Skin culture | Х | X | | | | X | X |
| Post surgical assessment | | | X | X | Х | х | Х |
| Blinded assessor to<br>evaluate for s/sx of<br>SSI | | | | | | | х |
| Assess for adverse events | X | X | X | X | X | х | х |
| medications | X | X | X | X | X | X | X |

<sup>&</sup>lt;sup>1</sup>Supplies will be given to participants at screening visit. Application will be done by the participant on the evening before surgery.

# References

- Abbey DM, Turner DM, Warson JS, Wirt TC, Scalley RD (1995) Treatment of postoperative wound infections following spinal fusion with instrumentation. J Spinal Disord 8:278–283CrossRefPubMed
- Balderston RA, Blumberg K (1991) Infection in spine surgery. In: Balderston RA, An HS (eds) Complications in spinal surgery. WB Saunders, Philadelphia, pp 157–168
- Glassman SD, Dimar JR, Puno RM, Johnson JR (1996) Salvage of instrumental lumbar fusions complicated by surgical wound infection. Spine 21:2163–2169CrossRefPubMed
- Keller RB, Pappas AM (1972) Infection after spinal fusion using internal fixation instrumentation. Orthop Clin North Am 3:99–111PubMed
- Kostuik JP, Israel J, Hall JE (1973) Scoliosis surgery in adults. Clin Orthop 93:225– 234CrossRefPubMed
- 6. Lonstein J, Winter R, Moe J, Gaines D (1973) Wound infection with Harrington instrumentation and spine fusion for scoliosis. Clin Orthop 96:222–233PubMed
- 7. Roberts FJ, Walsh A, Wing P, Dvorak M, Schweigel J (1998) The influence of surveillance methods on surgical wound infection rates in a tertiary care spinal surgery service. Spine 23:366–370CrossRefPubMed
- 8. West JL 3rd, Ogilvie JW, Bradford DS (1991) Complications of the variable screw plate pedicle screw fixation. Spine 16:576–579CrossRefPubMed
- Olsen MA, Mayfield J, Lauryssen C, Polish LB, Jones M, Vest J, Fraser VJ (2003) Risk factors for surgical site infection in spinal surgery. J Neurosurg Spine 98:149–155CrossRef
- Calderone RR, Garland DE, Capen DA, Oster H (1996) Cost of medical care for postoperative spinal infections. Orthop Clin North Am 27:171–182PubMed
- Davis H (1994) Increasing rates of cervical and lumbar spine surgery in the United States,
   1979–1990. Spine 19:1117–1123 (discussion 1123–1114) CrossRefPubMed
- 12. Tenney JH, Vlahov D, Salcman M, Ducker TB (1985) Wide variation in risk of wound infection following clean neurosurgery. Implications for perioperative antibiotic prophylaxis. J Neurosurg 62:243–247CrossRefPubMed
- 13. Klein JD, Hey LA, Yu CS, Klein BB, Coufal FJ, Young EP, Marshall LF, Garfin SR (1996) Perioperative nutrition and postoperative complications in patients undergoing spinal surgery. Spine 21:2676–2682CrossRefPubMed
- 14. Wimmer C, Gluch H, Franzreb M, Ogon M (1998) Predisposing factors for infection in spine surgery: a survey of 850 spinal procedures. J Spinal Disord 11:124–128PubMed

- Andreshak TG, An HS, Hall J, Stein B (1997) Lumbar spine surgery in the obese patient. J Spinal Disord 10:376–379CrossRefPubMed
- 16. Capen DA, Calderone RR, Green A (1996) Perioperative risk factors for wound infections after lower back fusions. Orthop Clin North Am 27:83–86PubMed
- 17. Patel N, Bagan B, Vadera S, Maltenfort MG, Deutsch H, Vaccaro AR, Harrop J, Sharan A, Ratliff JK (2007) Obesity and spine surgery: relation to perioperative complications. J Neurosurg Spine 6:291–297CrossRefPubMed
- Massie JB, Heller JG, Abitbol JJ, McPherson D, Garfin SR (1992) Postoperative posterior spinal wound infections. Clin Orthop Relat Res 284:99–108PubMed
- Simpson JM, Silveri CP, Balderston RA, Simeone FA, An HS (1993) The results of operations on the lumbar spine in patients who have diabetes mellitus. J Bone Joint Surg Am 75:1823–1829PubMed
- McPhee IB, Williams RP, Swanson CE (1998) Factors influencing wound healing after surgery for metastatic disease of the spine. Spine 23:726–732 (discussion 732– 733)CrossRefPubMed
- 21. Klein JD, Garfin SR (1996) Nutritional status in the patient with spinal infection. Orthop Clin North Am 27:33–36PubMed
- 22. Rechtine GR, Bono PL, Cahill D, Bolesta MJ, Chrin AM (2001) Postoperative wound infection after instrumentation of thoracic and lumbar fractures. J Orthop Trauma 15:566–569CrossRefPubMed
- Dahners LE, Mullis BH (2004) Effects of nonsteroidal anti-inflammatory drugs on bone formation and soft-tissue healing. J Am Acad Orthop Surg 12:139–143PubMed
- 24. Picada R, Winter RB, Lonstein JE, Denis F, Pinto MR, Smith MD, Perra JH (2000) Postoperative deep wound infection in adults after posterior lumbosacral spine fusion with instrumentation: incidence and management. J Spinal Disord 13:42—45CrossRefPubMed
- Borkhuu B, Borowski A, Shah SA, Littleton AG, Dabney KW, Miller F (2008) Antibioticloaded allograft decreases the rate of acute deep wound infection after spinal fusion in cerebral palsy. Spine 33:2300–2304CrossRefPubMed
- Dumitrescu CE, Collins MT (2008) McCune-Albright syndrome. Orphanet J Rare Dis 3:12CrossRefPubMed
- 27. Milbrandt TA, Johnston CE 2nd (2005) Down syndrome and scoliosis: a review of a 50-year experience at one institution. Spine 30:2051–2055CrossRefPubMed
- 28. Odent T, Accadbled F, Koureas G, Cournot M, Moine A, Diene G, Molinas C, Pinto G, Tauber M, Gomes B, de Gauzy JS, Glorion C (2008) Scoliosis in patients with Prader-Willi Syndrome. Pediatrics 122:e499–e503CrossRefPubMed

- 29. Tsirikos AI, Lipton G, Chang WN, Dabney KW, Miller F (2008) Surgical correction of scoliosis in pediatric patients with cerebral palsy using the unit rod instrumentation. Spine 33:1133–1140CrossRefPubMed
- Rihn JA, Lee JY, Ward WT (2008) Infection after the surgical treatment of adolescent idiopathic scoliosis: evaluation of the diagnosis, treatment, and impact on clinical outcomes.
   Spine 33:289–294CrossRefPubMed
- 31. Ho C, Sucato DJ, Richards BS (2007) Risk factors for the development of delayed infections following posterior spinal fusion and instrumentation in adolescent idiopathic scoliosis patients. Spine 32:2272–2277CrossRefPubMed
- 32. Sponseller PD, LaPorte DM, Hungerford MW, Eck K, Bridwell KH, Lenke LG (2000) Deep wound infections after neuromuscular scoliosis surgery: a multicenter study of risk factors and treatment outcomes. Spine 25:2461–2466CrossRefPubMed
- 33. Soultanis K, Mantelos G, Pagiatakis A, Soucacos PN (2003) Late infection in patients with scoliosis treated with spinal instrumentation. Clin Orthop Relat Res 411:116–123CrossRefPubMed
- 34. Li S, Zhang J, Li J, Lin J, Tian Y, Weng X, Qiu G (2002) Wound infection after scoliosis surgery: an analysis of 15 cases. Chin Med Sci J 17:193–198PubMed
- 35. Tsiodras S, Falagas ME (2006) Clinical assessment and medical treatment of spine infections. Clin Orthop Relat Res 444:38–50CrossRefPubMed
- 36. Pull ter Gunne AF, Cohen DB (2009) Incidence, prevalence and analysis of risk factors for surgical site infection following adult spinal surgery. Spine (in press)
- 37. Fang A, Hu SS, Endres N, Bradford DS (2005) Risk factors for infection after spinal surgery. Spine 30:1460–1465CrossRefPubMed
- 38. Eiselt, Debra (2009) Presurgical Skin Preparation With a Novel 2% Chlorhexidine Gluconate Cloth Reduces Rates of Surgical Site Infection in Orthopaedic Surgical Patients Orthopaedic Nursing: May/June 2009 Volume 28 Issue 3 p 141–145 doi: 10.1097/NOR.0b013e3181a469db
- 39. Karki S, Cheng AC. Impact of non-rinse skin cleansing with chlorhexidinegluconate on prevention of healthcare-associated infections and colonization with multi-resistant organisms: asystematic review. J Hosp Infect 2012;82:71e84.
- Climo MW, Yokoe DS, Warren DK, et al. Effect of daily chlorhexidinebathing on hospitalacquired infection. N Engl J Med 2013;368:533e542.
- 41. Milstone AM, Elward A, Song X, et al. Daily chlorhexidinebathing to reduce bacteraemia in critically ill children: a multicentre, cluster-randomised, crossover trial. Lancet 2013;381:1099e1106.

# Table of Contents:

- 1. Background and Significance
- 2. Hypothesis
- 3. Study Objectives
- 4. Methods
- 5. Patient Population
- 6. Enrollment
- 7. Inclusion/Exclusion Criteria
- 8. Data Collection
- 9. Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others:
- 10. Statistical Plan
- 11. Privacy/Confidentiality Issues
- 12. Follow-up and Record Retention

# 1. Background and Significance:

Surgical site infection (SSI) following spinal surgery is a frequent complication and results in higher morbidity, mortality and healthcare costs. SSI following adult spinal surgery is a frequent complication that has been reported to occur in 0.7–12.0% of patients and result in higher postoperative morbidity, mortality and health care costs. Vanderbilt University Medical Center SSI rate is 7%. Treatment for SSI can be challenging often requiring revision surgery, long-term antibiotics, and prolonged hospitalization. The accurate identification of risk factors is thus important in the development of strategies to prevent these potentially devastating infections.

The New CDC-definitions for surveillance of surgical site infections (1992) take into account 3 classes of surgical site infections (SSI): superficial incisional SSI, deep incisional SSI, and organ/space SSI. The most prevalent host-related risk factors for development of SSI are advanced age, morbid obesity, disease severity, an ASA score > 2, prolonged preoperative hospital stay, and infection at distal sites. Microbial contamination of the surgical site occurs mainly during the surgical intervention.

Although exogenous contamination from the surgical suite may be of concern, especially in clean operations, most surgical site infections are caused by microorganisms of the patient's own skin flora. SSI rates vary according to the type and duration of the surgical procedure. Proper surgical technique is probably the most important factor in the prevention of SSI. Modification of patient risk factors should be attempted whenever possible through use of

Modification of patient risk factors should be attempted whenever possible through use of adequate protocols for antimicrobial prophylaxis with antibiotics should be followed. Routine surveillance of surgical site infections is beneficial for SSI prevention and early detection. Additional prevention aimed at decreasing number of microorganisims on patient's skin preoperatively may decrease rates of SSI. Prior studies have reported daily use of 2% chlorhexidine gluconate (CHG) cloths has decreased rates of nosocomial bloodstream infections in those with central line catheters. Another study reported decreasing SSIs up to 50% when nursing staff instituted utilization of CHG cloths pre-op and daily post-op cleansing in-hospital. However, use of CHG cloths pre-operatively has not been routinely instituted. Many hospitals and service lines do not have a protocol for their use. Therefore study of such a population may prove worthy, as currently VUMC neuro-spine patients do not routinely utilize preoperative skin cleansing with CHG cloths.

This study proposes a randomized, controlled trial of neuro-spine patients of 2% chlorhexidine gluconate skin preparation cloths for the prevention of post op surgical site infections in spine patients.

# Hypothesis:

Use of CHG cloths the night before and morning of surgery (neckline to toes) will affect (decrease rates) of SSI compared to patients who receive routine standard of care (soap and water pre-op, day of surgery and daily post-operative).

# 3. Study Objectives:

- Randomize consented patients pre-operative to either study group (of 2% chlorhexidine gluconate cloths the night before and morning of surgery) or control (standard of care cleansing with soap and water) with follow-up through discharge for evaluation of SSI
- Evaluation for SSI development at 6 week (+/-) 1 week post-op visit.

 Measure change in skin flora by comparing skin swab cultures of those using the cloths and those who do not on day of surgery, post-op day 4 or hospital discharge and postop day 30

#### Methods:

Pre-operatively patients scheduled for neurosurgical spine cases will be evaluated and approached for interest, if consenting process completed, patients will be randomized to one of 2 arms in 1:1 through a block randomization table.

Those enrolled into the study arm will receive the CHG cloths and instructions for use from research personal. Those randomized to the control arm will receive standard of care skin cleansing by nursing staff.

All subjects who have signed consent will have a skin swab culture taken the day of screening and prior to cleansing with Chlorhexidine gluconate wipes close to the intended incision line. We will also obtain skin swab cultures at site of incision preoperatively on the day of surgery, post-op day 4 or time of discharge (which ever comes first) and at the 30 day follow up.

Both groups will be evaluated daily by study personnel for the development of SSI until postop day 4 or hospital discharge whichever one comes first.. Additional evaluations will take place at the 30 day (+/- 7 days) post-op visit. Blinded evaluators utilizing the CDC guideline will grade the incision line for presence of SSI. Measured change in skin flora will be performed by comparing skin swab cultures of intervention group versus standard of care group and individual changes pre and post operatively.

# 5. Patient Population:

Neurosurgical spine patients at Vanderbilt University Medical Center

#### 6. Enrollment:

170 patients will be enrolled.

# 7. Inclusion/Exclusion Criteria:

#### Inclusion Criteria

Patients scheduled for a neuro-spine procedure and have 2 of the following risk factors: Diabetic OR BMI>30 OR ASA>2 OR pre-operatively hospitalized OR >60 years old OR chronic steroids/immunosuppressive medications OR prior history of SSI

#### Exclusion Criteria

- 1) Unable to consent
- 2) Non English speaking
- 3) Known allergy to any of the ingredients contained in SAGE chlorhexidine gluconate cloths
- 4) Current infection or history of spine infections.
- 5) Patients with tumors or intradural spinal pathology.

# 8. Data Collection:

Data regarding demographics, health history and status, surgical course and hospitalization will be collected and entered into an electronic database. Patient data will be de-identified once entered into the database. Shared data will always be de-identified and accessed through Redcap, a secure web-based system.

# Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others:

Events determined by the Principal Investigator (PI) to be unanticipated problems involving risks to subjects will be reported by the PI or sub-investigator to the IRB within 10 working days of the Investigator's knowledge of the problem.

#### 10. Statistical Plan:

We are planning a study of independent cases and controls with 1 control(s) per case. Prior data indicate the rate of infection in the control group (those with risk factors, including superficial SSI) is 0.5, then just 150 evaluable subjects are needed to detect a 50% or greater reduction, with 80% power. We can also design a statistical analysis plan that uses the grade of SSI instead of binary yes/no to indicate presence of SSI. This should increase the power as well, for instance, if the SAGE cloths reduce the severity of (but does not completely prevent) infection in some patients.

# 11. Privacy/Confidentiality Issues

All reasonable efforts will be made to keep a patient's protected health information (PHI) private and confidential. There will be limited access to electronic medical records and deidentification of all records. Federal privacy guidelines will be followed when using or sharing any protected health information.

Data will be stored in Redcap, a secure web-based database conforming to the latest Vanderbilt IS security policies. Data from the study will be reported only in the aggregate.

Under the supervision of each site's PI, Vanderbilt research team members will view research records and collect data as identified above. Medical records will be stored separately from the data and remain on-site. All de-identified data-points will be entered directly into Redcap, a secure web-based database. No identified information will leave the site.

All study staff have completed employee education regarding patient confidentiality and have completed Human Subjects protection education (CITI course) as specified by the Vanderbilt IRB.

Through these interventions, we expect risks to privacy to be minimized.

# 12. Follow-up and Record Retention

Research Records will be retained by the Nursing Research Office for a period of six (6) years after the submission of the final report and close-out procedures on the research project for which the Research Records were prepared.

The retention of the original Research Records shall be the responsibilityNursing Research Office .

# Study Schema

| Procedure | screening | Day of surgery | POD 1 | POD 2 | POD 3 | POD4 or<br>discharge | 6 weeks<br>± 1 week<br>follow up<br>visit |
|---|---|---|---|---|---|---|---|
| Written informed consent | X | | | | | | |
| Medical history | Х | | | | | | |
| Urine pregnancy test | | Х | | | | | |
| BMI | х | | | | | | |
| Vital signs (HR, RR,<br>BP, T) | X | Х | X | X | X | x | Х |
| Randomization | Х | | | | | | |
| SAGE cloths for<br>treatment arm <sup>1</sup> | X | X | | | | | |
| Standard of care;<br>soap and water for<br>control arm | х | х | х | х | х | X | |
| Skin culture | Х | X | | | | X | X |
| Post surgical assessment | | | X | X | Х | х | Х |
| Blinded assessor to<br>evaluate for s/sx of<br>SSI | | | | | | | x |
| Assess for adverse events | X | X | X | X | X | X | X |
| medications | X | X | Х | X | Х | Х | X |

<sup>&</sup>lt;sup>1</sup>Supplies will be given to participants at screening visit. Application will be done by the participant on the evening before surgery.

# References

- Abbey DM, Turner DM, Warson JS, Wirt TC, Scalley RD (1995) Treatment of postoperative wound infections following spinal fusion with instrumentation. J Spinal Disord 8:278–283CrossRefPubMed
- Balderston RA, Blumberg K (1991) Infection in spine surgery. In: Balderston RA, An HS (eds) Complications in spinal surgery. WB Saunders, Philadelphia, pp 157–168
- Glassman SD, Dimar JR, Puno RM, Johnson JR (1996) Salvage of instrumental lumbar fusions complicated by surgical wound infection. Spine 21:2163–2169CrossRefPubMed
- Keller RB, Pappas AM (1972) Infection after spinal fusion using internal fixation instrumentation. Orthop Clin North Am 3:99–111PubMed
- Kostuik JP, Israel J, Hall JE (1973) Scoliosis surgery in adults. Clin Orthop 93:225– 234CrossRefPubMed
- 6. Lonstein J, Winter R, Moe J, Gaines D (1973) Wound infection with Harrington instrumentation and spine fusion for scoliosis. Clin Orthop 96:222–233PubMed
- 7. Roberts FJ, Walsh A, Wing P, Dvorak M, Schweigel J (1998) The influence of surveillance methods on surgical wound infection rates in a tertiary care spinal surgery service. Spine 23:366–370CrossRefPubMed
- 8. West JL 3rd, Ogilvie JW, Bradford DS (1991) Complications of the variable screw plate pedicle screw fixation. Spine 16:576–579CrossRefPubMed
- Olsen MA, Mayfield J, Lauryssen C, Polish LB, Jones M, Vest J, Fraser VJ (2003) Risk factors for surgical site infection in spinal surgery. J Neurosurg Spine 98:149–155CrossRef
- Calderone RR, Garland DE, Capen DA, Oster H (1996) Cost of medical care for postoperative spinal infections. Orthop Clin North Am 27:171–182PubMed
- Davis H (1994) Increasing rates of cervical and lumbar spine surgery in the United States,
   1979–1990. Spine 19:1117–1123 (discussion 1123–1114) CrossRefPubMed
- 12. Tenney JH, Vlahov D, Salcman M, Ducker TB (1985) Wide variation in risk of wound infection following clean neurosurgery. Implications for perioperative antibiotic prophylaxis. J Neurosurg 62:243–247CrossRefPubMed
- 13. Klein JD, Hey LA, Yu CS, Klein BB, Coufal FJ, Young EP, Marshall LF, Garfin SR (1996) Perioperative nutrition and postoperative complications in patients undergoing spinal surgery. Spine 21:2676–2682CrossRefPubMed
- 14. Wimmer C, Gluch H, Franzreb M, Ogon M (1998) Predisposing factors for infection in spine surgery: a survey of 850 spinal procedures. J Spinal Disord 11:124–128PubMed

- Andreshak TG, An HS, Hall J, Stein B (1997) Lumbar spine surgery in the obese patient. J Spinal Disord 10:376–379CrossRefPubMed
- 16. Capen DA, Calderone RR, Green A (1996) Perioperative risk factors for wound infections after lower back fusions. Orthop Clin North Am 27:83–86PubMed
- 17. Patel N, Bagan B, Vadera S, Maltenfort MG, Deutsch H, Vaccaro AR, Harrop J, Sharan A, Ratliff JK (2007) Obesity and spine surgery: relation to perioperative complications. J Neurosurg Spine 6:291–297CrossRefPubMed
- Massie JB, Heller JG, Abitbol JJ, McPherson D, Garfin SR (1992) Postoperative posterior spinal wound infections. Clin Orthop Relat Res 284:99–108PubMed
- Simpson JM, Silveri CP, Balderston RA, Simeone FA, An HS (1993) The results of operations on the lumbar spine in patients who have diabetes mellitus. J Bone Joint Surg Am 75:1823–1829PubMed
- McPhee IB, Williams RP, Swanson CE (1998) Factors influencing wound healing after surgery for metastatic disease of the spine. Spine 23:726–732 (discussion 732– 733)CrossRefPubMed
- 21. Klein JD, Garfin SR (1996) Nutritional status in the patient with spinal infection. Orthop Clin North Am 27:33–36PubMed
- 22. Rechtine GR, Bono PL, Cahill D, Bolesta MJ, Chrin AM (2001) Postoperative wound infection after instrumentation of thoracic and lumbar fractures. J Orthop Trauma 15:566–569CrossRefPubMed
- Dahners LE, Mullis BH (2004) Effects of nonsteroidal anti-inflammatory drugs on bone formation and soft-tissue healing. J Am Acad Orthop Surg 12:139–143PubMed
- 24. Picada R, Winter RB, Lonstein JE, Denis F, Pinto MR, Smith MD, Perra JH (2000) Postoperative deep wound infection in adults after posterior lumbosacral spine fusion with instrumentation: incidence and management. J Spinal Disord 13:42—45CrossRefPubMed
- 25. Borkhuu B, Borowski A, Shah SA, Littleton AG, Dabney KW, Miller F (2008) Antibiotic-loaded allograft decreases the rate of acute deep wound infection after spinal fusion in cerebral palsy. Spine 33:2300–2304CrossRefPubMed
- Dumitrescu CE, Collins MT (2008) McCune-Albright syndrome. Orphanet J Rare Dis 3:12CrossRefPubMed
- 27. Milbrandt TA, Johnston CE 2nd (2005) Down syndrome and scoliosis: a review of a 50-year experience at one institution. Spine 30:2051–2055CrossRefPubMed
- 28. Odent T, Accadbled F, Koureas G, Cournot M, Moine A, Diene G, Molinas C, Pinto G, Tauber M, Gomes B, de Gauzy JS, Glorion C (2008) Scoliosis in patients with Prader-Willi Syndrome. Pediatrics 122:e499–e503CrossRefPubMed

- 29. Tsirikos AI, Lipton G, Chang WN, Dabney KW, Miller F (2008) Surgical correction of scoliosis in pediatric patients with cerebral palsy using the unit rod instrumentation. Spine 33:1133–1140CrossRefPubMed
- 30. Rihn JA, Lee JY, Ward WT (2008) Infection after the surgical treatment of adolescent idiopathic scoliosis: evaluation of the diagnosis, treatment, and impact on clinical outcomes. Spine 33:289–294CrossRefPubMed
- 31. Ho C, Sucato DJ, Richards BS (2007) Risk factors for the development of delayed infections following posterior spinal fusion and instrumentation in adolescent idiopathic scoliosis patients. Spine 32:2272–2277CrossRefPubMed
- 32. Sponseller PD, LaPorte DM, Hungerford MW, Eck K, Bridwell KH, Lenke LG (2000) Deep wound infections after neuromuscular scoliosis surgery: a multicenter study of risk factors and treatment outcomes. Spine 25:2461–2466CrossRefPubMed
- Soultanis K, Mantelos G, Pagiatakis A, Soucacos PN (2003) Late infection in patients with scoliosis treated with spinal instrumentation. Clin Orthop Relat Res 411:116– 123CrossRefPubMed
- 34. Li S, Zhang J, Li J, Lin J, Tian Y, Weng X, Qiu G (2002) Wound infection after scoliosis surgery: an analysis of 15 cases. Chin Med Sci J 17:193–198PubMed
- 35. Tsiodras S, Falagas ME (2006) Clinical assessment and medical treatment of spine infections. Clin Orthop Relat Res 444:38–50CrossRefPubMed
- 36. Pull ter Gunne AF, Cohen DB (2009) Incidence, prevalence and analysis of risk factors for surgical site infection following adult spinal surgery. Spine (in press)
- 37. Fang A, Hu SS, Endres N, Bradford DS (2005) Risk factors for infection after spinal surgery. Spine 30:1460–1465CrossRefPubMed
- 38. Eiselt, Debra (2009) Presurgical Skin Preparation With a Novel 2% Chlorhexidine Gluconate Cloth Reduces Rates of Surgical Site Infection in Orthopaedic Surgical Patients Orthopaedic Nursing: May/June 2009 Volume 28 Issue 3 p 141–145 doi: 10.1097/NOR.0b013e3181a469db
- 39. Karki S, Cheng AC. Impact of non-rinse skin cleansing with chlorhexidinegluconate on prevention of healthcare-associated infections and colonization with multi-resistant organisms: asystematic review. J Hosp Infect 2012;82:71e84.
- 40. Climo MW, Yokoe DS, Warren DK, et al. Effect of daily chlorhexidinebathing on hospital-acquired infection. N Engl J Med 2013;368:533e542.
- 41. Milstone AM, Elward A, Song X, et al. Daily chlorhexidinebathing to reduce bacteraemia in critically ill children: a multicentre, cluster-randomised, crossover trial. Lancet 2013;381:1099e1106.